CLINICAL TRIAL: NCT03826680
Title: The Relationship of Modified Cormack Lehane Scores Between Preoperative Awake Flexible Fiberoptic Laryngoscopy and Intraoperative Direct Laryngoscopy in Thyroidectomies, a Prospective, Clinical Study
Brief Title: Modified Cormack Lehane Scores Evaluated by Laryngoscopy During Awake Versus Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr Cigdem Akyol Beyoğlu, Medical doctor, Istanbul University
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: 11/01/2019-6469
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Thyroid Cancer; Thyroid Nodule; Thyroid Adenoma
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible fiberoptic laryngoscopy (Active Comparator): Patients who will undergo thyroidectomy will be evaluated by an ENT physician by flexible fiberoptic laryngoscopy before the surgery
  Interventions: Procedure: Flexible fiberoptic laryngoscopy
- Direct laryngoscopy (Active Comparator): The same patients evaluated by flexible fiberoptic laryngoscopy will be evaluated by an anesthesiologist by direct laryngoscopy during surgery under general anesthesia
  Interventions: Procedure: Direct laryngoscopy

INTERVENTIONS:
Procedure: Flexible fiberoptic laryngoscopy — Patients who will undergo thyroidectomy will be evaluated by awake flexible fiberoptic laryngoscopy and during surgery by direct laryngoscopy under general anesthesia
  Arms: Flexible fiberoptic laryngoscopy
Procedure: Direct laryngoscopy — Patients who will undergo thyroidectomy evaluated before by ENT physician, will be evaluated by anesthesiologist in means of MCL score by direct laryngoscopy during surgery under general anesthesia
  Arms: Direct laryngoscopy

SUMMARY:
Nowadays, 5-step modified Cormack-Lehane scoring (MCL) system is frequently used in the observation of laryngeal structures by direct laryngoscopy.

Upper airways with flexible fiberoptic laryngoscopy are routinely evaluated in patients who are predicted to be difficult intubation, who have undergone head or neck surgery previously and who require vocal cords to be evaluated preoperatively. During this examination patients are awake; so the upper airway and the muscles in the base of the mouth have normal tonus and airway reflexes are active. When general anesthesia is applied to the same patients during direct laryngoscopy, the laryngeal view may not be as clear as awake flexible fiberoptic laryngoscopy, since a tonus loss occurs in the muscles after general anesthesia.

The aim of the study is to investigate the relationship between preoperative awake flexible fiberoptic laryngoscopy performed by ear- nose- throat (ENT) physicians in patients undergoing total thyroidectomy, and the MCL score during direct laryngoscopy after general anesthesia in the same patients. Thus, investigators would like to determine the reliability of airway evaluation with preoperative awake flexible fiberoptic laryngoscopy in predicting intubation conditions during tracheal intubation under general anesthesia.

DETAILED DESCRIPTION:
In daily practice, the upper airway evaluation is performed by the ENT physician with flexible fiberoptic laryngoscopy while the patients are awake one day before thyroidectomy. This evaluation will be done by the same ENT physician (EDG). Each patient will be kept in the neutral position and at the level of soft palate, the larynx will be observed by the flexible fiberoptic laryngoscopy and the laryngeal view and MCL score of these patients will be recorded.

The same patients will be taken to the preoperative care unit on the morning of operation and 20 G intravenous cannulation will be performed on the left hand. Patients' neck circumference and Mallampati score and presence of obstructive sleep apnea syndrome will be recorded. Patients will be taken to the operation theatre and standard monitoring will be performed consisting of electrocardiography (ECG), non-invasive blood pressure (BP) and peripheral O2 saturation. After induction of general anesthesia, the same anesthesiologist (CAB) will perform direct laryngoscopy by using Macintosh laryngoscope the MCL score will be recorded. The anesthesiologist will not know the MCL score that was previously evaluated by ENT physician during awake fiberoptic flexible laryngoscopy. Female and male patients will be intubated orotracheally with 7.5-8 internal diameter endotracheal tube, respectively. It will be recorded if the backward, upward, right, lateral pressure Maneuver (BURP) is applied during intubation. The maintenance of general anesthesia will be provided with 2% Sevoflurane in a 40% oxygen-air mixture.

After thyroidectomy is over patients will be extubated. The primary endpoint of the study was to evaluate the relationship between the MCL score, which was evaluated preoperatively, and the MCL score during direct laryngoscopy during intraoperative general anesthesia in awake patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo total or partial thyroidectomy
* American Society of Anesthesiologists class of I to III

Exclusion Criteria:

* Patients refusing to attend to study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Relation between MCL scores | 24 hours
  The primary outcome measure of the study is a 5 graded modified Cormack Lehane scores obtained from patients before and during thyroidectomy. The first measurement will be done one day before surgery, while patient is awake by flexible fiberoptic laryngoscopy. The second measurement will be done during surgery, after induction of general anesthesia by direct laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Guniz Koksal, Prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa Department of Anesthesiology, general surgery, ENT surgery, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
all collected individual participant data (IPD)